CLINICAL TRIAL: NCT02862301
Title: Epigenetic Evaluation of HAT/HDAC Activity in Peripheral Blood Mononuclear Cells From Patients With Clinically Isolated Syndrome and Analysis of the Relationship With the Pathophysiology and Disease Activity
Brief Title: Epigenetic Evaluation of HAT/HDAC Activity in PBMC From Patients With Clinically Isolated Syndrome
Acronym: EPIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: API/2015/64
Record Dates: First submitted 2016-08-03; First posted 2016-08-11 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Demyelinating Autoimmune Diseases, CNS
Keywords: Histone Deacetylases; Histone Acetyltransferases
MeSH Terms: conditions — Demyelinating Autoimmune Diseases, CNS | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Other): Healthy volunteers, free of any inflammatory disease. A blood sample is performed on the day of inclusion.
  Interventions: Biological: blood sample
- CIS group (Experimental): patients with Clinically isolated syndrome. A blood sample is performed on the day of inclusion and after 3 months.
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample

SUMMARY:
The aim of the study is to compare the enzymatic activity of HATs and HDACs in peripheral blood mononuclear cell (PBMC) of patients with a clinically isolated syndrome (CIS group) and healthy controls (control group).

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune inflammatory demyelinating disease of the central nervous system (CNS). Clinically isolated syndrome (CIS) is often a sign of multiple sclerosis and the term refers to the first episode of neurologic symptoms experienced by a patient. Possible presentations of CIS include optic neuritis, a brain stem and/or cerebellar syndrome, a spinal cord syndrome, or occasionally cerebral hemispheric dysfunction. An accurate diagnosis at this time is important because people with a high risk of developing MS are encouraged to begin treatment in order to delay or prevent a second neurologic episode and, therefore, the onset of MS.

The innate and adaptative immune systems play an important role in pathophysiology of MS, acting in interaction with environmental, genetic, and epigenetic factors.

Epigenetic modifications, such as DNA methylation and histone modification, alter DNA accessibility and chromatin structure, thereby regulating patterns of gene expression. These processes are crucial to normal development and differentiation of distinct cell lineages in the adult organism. Histone acetylation, through the family of histone acetyl transferase (HAT), is most consistently associated with promoting transcription. Deacetylation of histones correlates with CpG methylation and the inactive state of chromatin. There are 4 classes of histone deacetylase enzymes (HDACs), with members capable of deacetylation of histones and/or other protein targets. Acetylation homeostasis is a key regulator of both immune cell activation. Of note, potent histone deacetylase inhibitors (HDACi) endowed with antiinflammatory and neuroprotective properties have been identified. Efficacy of HDACi in experimental models of MS has been reported consistently. This study could provide information on the mechanisms involved.

ELIGIBILITY:
Inclusion Criteria:

* Clinically isolated syndrome within the last 6 weeks (CIS group)
* Healthy volunteer, free of any inflammatory disease (control group)
* Patient able to understand the reason of the study
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Systemic corticosteroid therapy (>1mg/kg)
* Immunosuppressive/immunomodulatory therapy (prior or ongoing) (CIS group)
* Patient with ongoing infection (Control group)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
HDAC/ HAT enzymatic activity (ratio) | day of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Béreau, MD, Principal Investigator — CHU de Besançon
Locations (1):
- University Hospital, Besançon, France

IPD SHARING:
Plan to Share IPD: No